CLINICAL TRIAL: NCT02671357
Title: Enhanced Recovery After Minimally Invasive Pancreaticoduodenectomy With Stented Pancreaticogastrostomy and Roux-en-y Gastro-enterostomy
Brief Title: Enhanced Recovery After Minimally Invasive Pancreaticoduodenectomy
Acronym: ERAMIP
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Baki Topal, Professor, Doctor, University Hospital, Gasthuisberg
Other Study IDs: ERAMIP
Record Dates: First submitted 2016-01-22; First posted 2016-02-02 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Neoplasms; Periampullary Neoplasms
Keywords: pancreatic surgery; neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ERAMIP with EEN: Minimally invasive pancreaticoduodenectomy (MIPD) with stented pancreatic-gastrostomy & Roux-en-Y reconstruction of the biliary limb of the hepatico-jejunostomy onto the efferent limb of the gastro-enterostomy (RY-GES). All patients are submitted to an ERAS trajectory with EEN
  Interventions: Procedure: ERAMIP

INTERVENTIONS:
Procedure: ERAMIP — 3D-LPD with stented umbrella-pancreaticogastrostomy & Roux-en-Y reconstruction of the biliary limb of the hepatico-jejunostomy onto the efferent limb of the gastro-enterostomy (RY-GES)

SUMMARY:
This prospective observational cohort study aims to improve the postoperative course after minimally invasive pancreaticoduodenectomy (MIP) with stented pancreaticogastrostomy (sPG) for pancreatic head or peri-ampullary neoplasms. Patients are submitted to an enhanced recovery after surgery (ERAS) program with early enteral nutrition (EEN).

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is the standard of care for patients with malignant or benign disease of the pancreatic head or peri-ampullary region. The postoperative course after PD is strongly dependent of the occurrence of pancreatic fistula (POPF) and/or delayed gastric emptying (DGE). In a recent multicentre randomized controlled trial, the investigators have shown pancreaticogastrostomy (PG; without a stent in the pancreatic duct) to be associated with 8% POPF rate, significantly lower than pancreaticojejunostomy (20%) (1). Since then, PG reconstruction is considered the standard of care in PD, which is also underlined in more recent systematic reviews.

In patients without POPF after PD, the length of hospital stay is determined by the occurrence of DGE, which is poorly understood and currently lacks any effective treatment. Patients who developed DGE after PD with PG anastomosis (n=18; 20%) had a significantly (p=0.014) longer (mean + sem) length of hospital stay (LOS) of 26.3 + 1.58 days, as compared to 22.4 + 1.27 days for patients without DGE (n=69). These figures are observed in the investigators' center as part of the multicentre RCT.

Enhanced recovery after surgery (ERAS) or fast-track (FT) programs are able to reduce postoperative length of hospital stay (LOS). Indeed recently, ERAS or FT programs have been implemented successfully in PD (2). Patients were discharged 4 days earlier in the ERAS group, without a negative effect on the clinical outcome. Still, many surgeons are reluctant to implement ERAS programs because they fear compromising patient safety.

In efforts to improve the outcomes of PD, many surgical techniques have been evaluated to restore the pancreatic digestive continuity after PD. However, the best way to ensure this and whether or not to perform the procedure via standard open or minimally invasive, i.e. 2- or 3-dimensional laparoscopic (3D-LPD) or 3-dimensional robotic surgery (RPD), is still under debate. The investigators have passed the learning curve of 50 3D-LPD and hypothesize the implementation of ERAS and EEN in 3D-LPD can improve short-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, who undergo MIP + sPG for a pancreatic or peri-ampullary tumor
* Patients with and without pre-operative biliary drainage (for obstructive jaundice)
* Patients fit for minimally invasive pancreaticoduodenectomy (MIP)
* Informed consent signed

Exclusion Criteria:

* Pregnancy
* MIP for pancreatic trauma
* MIP for complications of endoscopic retrograde cholangio-pancreaticography (ERCP)
* Reconstruction of the portal vein or superior mesenteric vein
* Any arterial reconstruction at the time of surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic or peri-ampullarf neoplasms to undergo minimally invasive pancreaticoduodenectomy
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
The incidence of severe complications | From date of pancreaticoduodenectomy until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 3 months
  Severe complications are classified according to the Clavien-Dindo Classification, i.e. Therapy Oriented Severity Grading Score of postoperative complications (TOSGS grade 3 or more): complication that needs interventional therapy under local or general anaesthesia

SECONDARY OUTCOMES:
Postoperative in-hospital, 30-day and 90-day mortality | From date of pancreaticoduodenectomy until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 3 month
  Postoperative mortality rate

OTHER OUTCOMES:
Clinical postoperative pancreatic fistula (POPF) rate | From date of pancreaticoduodenectomy until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 3 months
  The incidence of POPF will be registered and defined according to the ISGPF
Postoperative bleeding (PPH) rate | From date of discharge from hospital until date of re-admission to hospital within 2 weeks after discharge, assessed up to 3 months
  The incidence of PPH will be registered and defined according to the ISGPF
Length of postoperative hospital stay (LOS) | From date of pancreaticoduodenectomy until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 3 months. Readmissions within 30days after discharge will be added to the duration of LOS.
  Length of hospital stay (days) will be registered starting from the day of surgery until discharge
Delayed gastric emptying (DGE) rate | From date of pancreaticoduodenectomy until the date of discharge from hospital or date of death from any cause, whichever came first, assessed up to 3 months
  The incidence of DGE will be registered and defined according to the ISGPF

CONTACTS AND LOCATIONS:
Overall Officials: Baki Topal, MD, PhD, Principal Investigator — University Hospitals KU Leuven
Locations (1):
- University Hospitals KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Topal B, Fieuws S, Aerts R, Weerts J, Feryn T, Roeyen G, Bertrand C, Hubert C, Janssens M, Closset J; Belgian Section of Hepatobiliary and Pancreatic Surgery. Pancreaticojejunostomy versus pancreaticogastrostomy reconstruction after pancreaticoduodenectomy for pancreatic or periampullary tumours: a multicentre randomised trial. Lancet Oncol. 2013 Jun;14(7):655-62. doi: 10.1016/S1470-2045(13)70126-8. Epub 2013 May 2. PMID 23643139
- [Background] Williamsson C, Karlsson N, Sturesson C, Lindell G, Andersson R, Tingstedt B. Impact of a fast-track surgery programme for pancreaticoduodenectomy. Br J Surg. 2015 Aug;102(9):1133-41. doi: 10.1002/bjs.9856. Epub 2015 Jun 4. PMID 26042725
- [Derived] Topal H, Jaekers J, Geers J, Topal B. Prospective cohort study on short-term outcomes of 3D-laparoscopic pancreaticoduodenectomy with stented pancreaticogastrostomy. Surg Endosc. 2023 Feb;37(2):1203-1212. doi: 10.1007/s00464-022-09609-9. Epub 2022 Sep 26. PMID 36163561